CLINICAL TRIAL: NCT04604366
Title: Comparison of Vaginal Versus Sublingual Misoprostol in the Treatment of First Trimester Missed Miscarriage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Islamabad Medical and Dental College (Other)
Responsible Party: Principal Investigator, Afnan Rizwan, Assistant professor, Islamabad Medical and Dental College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IslamabadMDC
Record Dates: First submitted 2020-10-06; First posted 2020-10-27 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Miscarriage; Misoprostol
Keywords: mesoprostol; vaginal; sublingual
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Misoprostol; Alprostadil

STUDY DESIGN:
Who Masked: Participant
Masking Description: lottery method will be used .one hundred and twenty slips will be made .60 will be marked as group A and 60 will be as Group B. these will be put in basket .and will be picked by the team member
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vaginal mesoprostol (Active Comparator): Vaginal dose---800 microgram 3 hourly two doses
  Interventions: Drug: misoprostol
- sublingual mesoprostol (Experimental): Sub lingual 600 microgram 3 hourly two doses
  Interventions: Drug: misoprostol

INTERVENTIONS:
Drug: misoprostol — it stimulates uterine contractions
  Other Names: prostaglandin E1

SUMMARY:
The miscarriage is one of the adverse outcomes of pregnancy and is responsible for stress and anxiety of the couple. there are different types of miscarriages.missed miscarriage also known as early fetal demise is one of the type of miscarriage in which patient is mostly asymptomatic but Ultrasound shows absent fetal cardiac activity.Traditionally surgical evacuation of uterus was the treatment of choice for miscarriage.The treatment of miscarriage has evolved significantly in recent years.medical management using misoprostol is the newest treatment option.Misoprostol is a synthetic prostaglandin E(1) analogue that is commonly used for medical miscarriage It can be given orally, vaginally and sublingually.

DETAILED DESCRIPTION:
This study will be conducted in gynae and obstetric department of Akbar Niazi teaching hospital.Patients coming to gynaecology Outpatient department having confirmed diagnosis of missed miscarriage on pelvic ultrasound in first trimester will be enrolled after taking written consent for medical treatment.Patients will be randomly selected for oral or vaginal route of misoprostol,dosage according to international federation of gynaecology and obstetrics protocol.

Vaginal dose---800 microgram 3 hourly two doses Sub lingual 600 microgram 3 hourly two doses Patients will be observed for vaginal bleeding and expulsion for 24 hours if no expulsion or vaginal bleeding occurred then dose will be repeated .maximum of two cycles will be given. Failure of treatment confirmed by Ultrasonography will be dealt with surgical evacuation In case of heavy vaginal bleeding or expulsion pelvic USG will be done to confirm.After admission baseline investigation and coagulation studies will be performed . demographic details will be recorded...

Patients will be assessed for time taken in complete expulsion of conceptus. No of doses required Need for surgical evacuation Haemorrhage Fall in Hb level Need of blod transfusion Patient satisfaction Side effects of misoprostol like shivering,fever diarrhea and oral ulcers and others EXCLUSION CRITERIA patients who opted for surgical management or expectant management. Gestational age >13 weeks Patients with co-morbidity

Sample size: A total of 120 women will be selected for the study, divided into two equal groups of 60 women in each group. The sample size was calculated by WHO sample size calculator with of help of 5% level of significance, 90% power of test, 48% vs. 20% overall complication rate in sub inguinal and vaginal misoprostol groups (???).

Statistical analysis: All the collected data will be entered into SPSS v. 21 for analysis. Quantitative data will be presented in the form of mean ± standard deviation. Independent sample t-test will be applied to compare the quantitative variables (like age and gestational age) between both groups. Frequency with percentages will be calculated for qualitative data and chi-square test will be used to compare the qualitative variables (like abortion and complications) between both groups. P-value ≤ 0.05 will be taken as significant.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of missed miscarriage on pelvic ultrasound
* Gestational age ≤ 13 weeks

Exclusion Criteria:

* Patients who opted for surgical or expectant management.
* Patients with co-morbidity

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with complete expulsion of conceptus. | six months
  primary outcome measure is to record the number of patients in each group who achieved complete expulsion of products of conception.complete expulsion will be confirmed by pelvic USG

SECONDARY OUTCOMES:
Number of patients having side effects of misoprostol like shivering, fever diarrhea and oral ulcers and others | six months
  through physical examination and detailed history

CONTACTS AND LOCATIONS:
Locations (1):
- Islamabad Medical and Dental College, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dehbashi Z, Moosazadeh M, Afshari M. COMPARISON BETWEEN SUBLINGUAL AND VAGINAL ROUTE OF MISOPROSTOL IN MANAGEMENT OF FIRST TRIMESTER MISCARRIAGE MISSING. Mater Sociomed. 2016 Jul 24;28(4):271-273. doi: 10.5455/msm.2016.28.271-273. PMID 27698600